CLINICAL TRIAL: NCT02073084
Title: A Thorough Corrected QT Interval Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: K-877-102
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Sequence A (Other): Sequence A
  Interventions: Drug: K-877 Low Dose; Drug: Moxifloxacin; Other: Placebo; Drug: K-877 High Dose
- Sequence B (Other): Sequence B
  Interventions: Drug: K-877 Low Dose; Drug: Moxifloxacin; Other: Placebo; Drug: K-877 High Dose
- Sequence C (Other): Sequence C
  Interventions: Drug: K-877 Low Dose; Drug: Moxifloxacin; Other: Placebo; Drug: K-877 High Dose
- Sequence D (Other): Sequence D
  Interventions: Drug: K-877 Low Dose; Drug: Moxifloxacin; Other: Placebo; Drug: K-877 High Dose

INTERVENTIONS:
Drug: K-877 Low Dose — K-877 Low Dose
Drug: Moxifloxacin
Other: Placebo
Drug: K-877 High Dose — K-877 High Dose

SUMMARY:
The purpose of this study is to determine the effects of K-877 on ECG parameters with a focus on cardiac repolarization compared with placebo in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study specific evaluation is performed.
* Subject is a healthy adult male or female volunteer, of any race and ethnicity, between the ages of 18 and 45 years, inclusive.
* Subject has a body mass index of 18 to 30 kg/m2, inclusive.

Exclusion Criteria:

* Subject has clinically relevant abnormalities in the screening or check in assessments.
* Subject has a supine blood pressure after resting for at least 5 minutes that is higher than 140 mm Hg systolic or 90 mm Hg diastolic, or lower than 90 mm Hg systolic or 60 mm Hg diastolic.
* Subject has a supine Heart Rate (HR) (as measured at Screening or Check-in during collection of vital signs) after resting for at least 5 minutes that is outside the range of 40 to 90 beats per minute.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
QTcI (QT interval corrected) duration | 24 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States